CLINICAL TRIAL: NCT05790720
Title: Development of a Pharmacodynamic Model for Propofol in Older Adults (Development phaRmacodynamic mOdel Propofol oLdEr adulTs: DROPLET)
Brief Title: Development of a Pharmacodynamic Model for Propofol in Older Adults
Acronym: DROPLET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 230125002
Record Dates: First submitted 2023-03-02; First posted 2023-03-30 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-05

CONDITIONS: Aged
Keywords: Propofol; TCI; TIVA
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Pharmacokinetic-pharmacodynamic model that uses the pharmacokinetic parameters of the Eleveld model and new pharmacodynamic parameters derived from frontal EEG in a population older than 65 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Patients older than 65 years of age will receive an intravenous infusion of Propofol with prespecified plasma targets. During its administration, registration of BIS values, frontal electroencephalography, and clinical signs of consciousness will be performed. Two models will be created and compared retrospectively: BIS (Eleveld Validation) and EEG Frontal Marker (New model).
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Patients older than 65 years of age will receive an intravenous infusion of Propofol with prespecified plasma targets. During its administration, registration of BIS values, frontal electroencephalography, and clinical signs of consciousness will be performed.

SUMMARY:
The goal of this pharmacodynamic study is to develop a model for Propofol administration for older adults (>65 years). The main objective is to create a model based on a new pharmacodynamic parameter, derived from frontal electroencephalogram (EEG), to admininster Propofol in older adults. With this new model, the investigators aim to:

* Evaluate the relationship between the plasmatic concentration, described by the Eleveld pharmacokinetic model, versus the effect of the drug represented with a new parameter derived from the intraoperative frontal EEG.
* To validate the predictive ability of Eleveld's pharmacokinetic-pharmacodynamic model, based on the bispectral index (BIS), compared to the new model based on a parameter derived from intraoperative frontal EEG.

Participants will be asked to answer preoperative questionnaires, receive a Propofol intravenous infusion concomitantly with continuous BIS and EEG monitoring, and to be evaluated for clinical sings of loss and return of consciousness.

DETAILED DESCRIPTION:
The administration of intravenous anesthetics in the elderly population requires adequate titration to avoid deleterious effects derived from overdosing or underdosing. Older patients show greater sensitivity to similar doses of propofol compared to younger patients. In addition, there is extensive interindividual variability among older patients, which would also explain the different responses to the same dose of drugs. This variability would be secondary to differences in comorbidities and physiological age, in contrast to chronological age, which would not explain the differences found in response to anesthetics in these patients.

One way in which an attempt has been made to make the doses of anesthetics in different patients comparable is the use of models that predict what infusion rate is required to maintain a given concentration at the site of drug action. The relationship between a propofol effect site concentration (Ce) with a given effect can be represented by pharmacodynamic (PD) models. Recently, Eleveld et al. created a pharmacokinetic-pharmacodynamic (PKPD) model for the administration of intravenous propofol in a population of wide ages, including neonates to older patients. However, the pharmacodynamic parameter used in this model was the BIS index, which has been questioned for its use in older adults. In addition, the creation of this PD model only included 3 patients older than 70 years, so the underrepresentation of this age group in the construction of the model could affect its performance, making it even more difficult to correctly predict the effect in this population.

Anesthetic drugs exert their desired hypnotic effect on the brain. Brain electrical activity can be monitored non-invasively by recording electrical potential on the cranial surface using electrodes. The electroencephalographic (EEG) changes observed with the administration of anesthetics are usually systematic across different patients. These have been described and have been used to identify different phases of anesthetic "depth" or hypnosis. In addition, the representation of the EEG signal by means of a spectrogram has facilitated the incorporation of this information into commercial EEG monitors that previously only included highly processed indices such as the BIS.

Within the EEG patterns of the spectrogram described for anesthetic maintenance with propofol, the alpha (8-12 Hz) and delta (1-4 Hz) oscillations stand out. However, the power of alpha oscillations decreases with age and with other changes that are associated with age, such as decreased cognitive ability, increased comorbidities and brain vulnerability. Therefore, guiding our administration of propofol based on obtaining a pattern of alpha predominance appears to be difficult in this aged population.

The general objective of this work is to build a PKPD model that uses the pharmacokinetic parameters of the Eleveld model and new pharmacodynamic parameters derived from the frontal EEG in a population older than 65 years. Our hypothesis is that the Eleveld PKPD model, modified with this new pharmacodynamic parameter, will predict better the hypnotic effect of propofol than the original Eleveld PKPD model, in adult patients older than 65 years.

The creation of a PKPD model of propofol for the population over 65 years of age would allow a better titration of this drug to avoid possible deleterious effects secondary to its under or overdosage.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non-cardiac elective surgery requiring general anesthesia
* American Society of Anesthesiologists Physical Status I to III

Exclusion Criteria:

* Patients undergoing emergency surgery
* Neurosurgical patients
* History of alcohol abuse or recreational drug use
* Known allergie to Propofol
* Body mass index ≥ 35 Kg m-2
* Unstable heart failure

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Performance Error (PE) | Intravenous infusion start to one minute after start of burst suppression in EEG
  Difference between the measured (according to Eleveld) and predicted concentrations, divided by the predicted concentration. Multiplied by 100. Unit of measure: percentage (%).

SECONDARY OUTCOMES:
Median Absolute Performance Error (MDAPE) | Intravenous infusion start to one minute after start of burst suppression in EEG
  Median Absolute Performance Error (MDAPE) is the median PE and is a measure of how close the predicted concentration is to the measured concentration (Accuracy). Unit of measure: percentage (%).
Median Prediction Error (MDPE) | Intravenous infusion start to one minute after start of burst suppression in EEG
  Median Prediction Error (MDPE) is a measure of the overall bias of the predictions; it indicates whether the model systematically overshoots or undershoots the target. Unit of measure: percentage (%).
Time of Loss of response (LOR) | Intravenous infusion start to one minute after start of burst suppression in EEG
  Loss of response (LOR) is defined as the time when patients stop responding to verbal commands, light tactile stimulation, and the eyelid reflex. Unit of measure: time (seconds).
Time of Burst-suppression (BS) | Intravenous infusion start to one minute after start of burst suppression in EEG
  Burst-suppression (BS) consists of alternating episodes of isoelectric flat EEG periods with bursts of slow waves, including systemic and quasiperiodic variation where high voltage and isoelectric periods have variations between and within bursts. Unit of measure: time (seconds).
Time of Return of response (ROR). | Intravenous infusion start to one minute after start of burst suppression in EEG
  Return of response (ROR) is defined as the response to verbal stimulation and mild tactile stimulation. Unit of measure: time (seconds).

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schnider TW, Minto CF, Shafer SL, Gambus PL, Andresen C, Goodale DB, Youngs EJ. The influence of age on propofol pharmacodynamics. Anesthesiology. 1999 Jun;90(6):1502-16. doi: 10.1097/00000542-199906000-00003. PMID 10360845
- [Background] Andres TM, McGrane T, McEvoy MD, Allen BFS. Geriatric Pharmacology: An Update. Anesthesiol Clin. 2019 Sep;37(3):475-492. doi: 10.1016/j.anclin.2019.04.007. Epub 2019 Jun 19. PMID 31337479
- [Background] Vuyk J. Pharmacodynamics in the elderly. Best Pract Res Clin Anaesthesiol. 2003 Jun;17(2):207-18. doi: 10.1016/s1521-6896(03)00008-9. PMID 12817915
- [Background] Roy RC. Choosing general versus regional anesthesia for the elderly. Anesthesiol Clin North Am. 2000 Mar;18(1):91-104, vii. doi: 10.1016/s0889-8537(05)70151-6. PMID 10935002
- [Background] Warner MA, Saletel RA, Schroeder DR, Warner DO, Offord KP, Gray DT. Outcomes of anesthesia and surgery in people 100 years of age and older. J Am Geriatr Soc. 1998 Aug;46(8):988-93. doi: 10.1111/j.1532-5415.1998.tb02754.x. PMID 9706888
- [Background] Eleveld DJ, Colin P, Absalom AR, Struys MMRF. Pharmacokinetic-pharmacodynamic model for propofol for broad application in anaesthesia and sedation. Br J Anaesth. 2018 May;120(5):942-959. doi: 10.1016/j.bja.2018.01.018. Epub 2018 Mar 12. PMID 29661412
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Kim MC, Fricchione GL, Brown EN, Akeju O. Role of electroencephalogram oscillations and the spectrogram in monitoring anaesthesia. BJA Educ. 2020 May;20(5):166-172. doi: 10.1016/j.bjae.2020.01.004. Epub 2020 Feb 20. No abstract available. PMID 33456946
- [Background] Purdon PL, Pierce ET, Mukamel EA, Prerau MJ, Walsh JL, Wong KF, Salazar-Gomez AF, Harrell PG, Sampson AL, Cimenser A, Ching S, Kopell NJ, Tavares-Stoeckel C, Habeeb K, Merhar R, Brown EN. Electroencephalogram signatures of loss and recovery of consciousness from propofol. Proc Natl Acad Sci U S A. 2013 Mar 19;110(12):E1142-51. doi: 10.1073/pnas.1221180110. Epub 2013 Mar 4. PMID 23487781
- [Background] Purdon PL, Pavone KJ, Akeju O, Smith AC, Sampson AL, Lee J, Zhou DW, Solt K, Brown EN. The Ageing Brain: Age-dependent changes in the electroencephalogram during propofol and sevoflurane general anaesthesia. Br J Anaesth. 2015 Jul;115 Suppl 1(Suppl 1):i46-i57. doi: 10.1093/bja/aev213. PMID 26174300
- [Background] Giattino CM, Gardner JE, Sbahi FM, Roberts KC, Cooter M, Moretti E, Browndyke JN, Mathew JP, Woldorff MG, Berger M; MADCO-PC Investigators. Intraoperative Frontal Alpha-Band Power Correlates with Preoperative Neurocognitive Function in Older Adults. Front Syst Neurosci. 2017 May 8;11:24. doi: 10.3389/fnsys.2017.00024. eCollection 2017. PMID 28533746
- [Background] Touchard C, Cartailler J, Leve C, Serrano J, Sabbagh D, Manquat E, Joachim J, Mateo J, Gayat E, Engemann D, Vallee F. Propofol Requirement and EEG Alpha Band Power During General Anesthesia Provide Complementary Views on Preoperative Cognitive Decline. Front Aging Neurosci. 2020 Nov 27;12:593320. doi: 10.3389/fnagi.2020.593320. eCollection 2020. PMID 33328973
- [Background] Kaiser HA, Hirschi T, Sleigh C, Reineke D, Hartwich V, Stucki M, Rummel C, Sleigh J, Hight D. Comorbidity-dependent changes in alpha and broadband electroencephalogram power during general anaesthesia for cardiac surgery. Br J Anaesth. 2020 Oct;125(4):456-465. doi: 10.1016/j.bja.2020.06.054. Epub 2020 Jul 31. PMID 32747077
- [Background] Shao YR, Kahali P, Houle TT, Deng H, Colvin C, Dickerson BC, Brown EN, Purdon PL. Low Frontal Alpha Power Is Associated With the Propensity for Burst Suppression: An Electroencephalogram Phenotype for a "Vulnerable Brain". Anesth Analg. 2020 Nov;131(5):1529-1539. doi: 10.1213/ANE.0000000000004781. PMID 33079876